CLINICAL TRIAL: NCT01362556
Title: Blood Gas Analysis and Buffering In Cardiac Arrest - A Multicenter, Prospective, Randomised, Double Blind Prehospital Trial to Evaluate the Impact of Early Blood-gas-analysis Targeted Buffer Therapy on ROSC After OOHCA
Brief Title: Blood Gas Analysis and Buffering In Cardiac Arrest
Acronym: BABICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Prause Gerhard, MD, Prof Dr, Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BABICA
Record Dates: First submitted 2011-04-27; First posted 2011-05-30 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-06

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Sodium Bicarbonate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium Chloride (Placebo Comparator): Group receiving sodium chloride 0.9% after arterial blood gas analysis in cardiac arrest.
  Interventions: Drug: Sodium Chloride
- Sodium Bicarbonate (Active Comparator): Group receiving targeted sodium bicarbonate 8% therapy after arterial blood gas analysis in cardiac arrest.
  Interventions: Drug: Sodium bicarbonate

INTERVENTIONS:
Drug: Sodium bicarbonate — Administration of a calculated amount of sodium bicarbonate 8% [SB] after arterial blood gas measurement according to Base Excess [BE] and Body weight [kg].
  Formula: SB [ml] = -BE * kg * 0.1
  Arms: Sodium Bicarbonate
Drug: Sodium Chloride — Administration of a calculated amount of sodium chloride 0.9% [SC] after arterial blood gas measurement according to Base Excess [BE] and Body weight [kg].
  Formula: SC [ml] = -BE * kg * 0.1
  Arms: Sodium Chloride

SUMMARY:
The debate over the administration of sodium bicarbonate in cardiac arrest has been going on for several decades, swinging like a pendulum from "first-line drug" to "not indicated" to the recent guidelines advocating "a small bolus under special conditions (metabolic acidosis, intoxication, long-term resuscitation)". A targeted, blood-gas controlled application under optimised ventilation conditions has not yet been evaluated prehospitally. Our preliminary studies have shown that an arterial puncture/line as well as measurement of blood gases is feasible in preclinical conditions. This multicentre trial including 5 centres and 10 physician-staffed emergency systems is designed to compare, in a prospective randomised controlled study, the effect of a calculated dosage of sodium bicarbonate based on the patient´s base deficit and weight, on ROSC (= return of spontaneous circulation) and on the secondary survival of cardiac arrest patients. The null hypothesis is that there is no or negative impact on survival.

ELIGIBILITY:
Inclusion Criteria:

* prehospitally started cardiopulmonary resuscitation (CPR)
* advanced cardiac life support provided
* age >18 years
* arterial pH < 7,2
* arterial BE < -12
* arterial pCO2 15-75 mmHg
* arterial pO2 >35 mmHg

Exclusion Criteria:

* women of childbearing age
* traumatic cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Rate of return of spontaneous circulation (ROSC) | Within five hours from start of resuscitation.

SECONDARY OUTCOMES:
Survival to discharge after cardiac arrest | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
  Discharge from hospital
Survival after one year of hospital discharge | One year after event

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Prause, Prof. Dr., Principal Investigator — Medical University of Graz
Locations (6):
- Austria (6):
  - Landeskrankenhaus Klagenfurt, Klagenfurt, Carinthia
  - Landesklinikum Wiener Neustadt, Wiener Neustadt, Lower Austria
  - Landeskrankenhaus Bruck / Mur, Bruck / Mur, Styria
  - LKH Graz West, Graz, Styria
  - Medical University Graz, Graz, Styria
  - AKH Linz, Linz, Upper Austria